CLINICAL TRIAL: NCT03419949
Title: Comparison of Oral Lamotrigine Versus Pregabalin for Control of Acute and Chronic Pain Following Modified Radical Mastectomy: Controlled Double-blind Study
Brief Title: Comparison of Oral Lamotrigine Versus Pregabalin for Control of Acute and Chronic Pain
Status: Available | Type: Expanded Access
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma elkomy, principal investigator, Assiut University
Other Study IDs: Comparison of oral lamotrigine
Record Dates: First submitted 2018-01-27; First posted 2018-02-05 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Acute and Chronic Pain Following Modified Radical Mastectomy
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Lamotrigine; Pregabalin

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: oral lamotrigine 100 mg — Pain relief drug Lamotrigine inhibits the voltage-gated sodium and calcium channels. Inhibition of the voltage-gated sodium channel stabilizes the presynaptic neuronal membrane, thus preventing the release of excitatory neurotransmitters such as glutamate and inhibiting sustained repetitive neuronal firing
  Other Names: lamictal
Drug: oral pregabalin 150 mg — Pain relief using drug Pregabalin is a structural analogue of the inhibitory neurotransmitter gama-aminobutyric acid (GABA), with anticonvulsant, antihyperalgesic, and anxiolytic properties
  Other Names: lyrica

SUMMARY:
Breast cancer is the most frequent neoplastic tumor in women, and surgical treatment is indicated in most patients. Complications related to this treatment, such as post-mastectomy pain syndrome (PMPS), a persistent pain that develops after surgery, have been reported. Although the genesis of the pain is multifactorial, sectioning of the intercostobrachial nerve is the nerve lesion diagnosed more often (1) ..

Pain relief using drugs with high efficacy provides significant improvement in the patients' lives. Drugs like lamotrigine (LTG) and gabapentin (GBP) have the ability to overcome the symptoms of neuropathic pain (4).

Both LTG and PGB have been extensively reviewed in the past for management of painful neuropathic conditions (5)

DETAILED DESCRIPTION:
This study will be carried out after being approved from the Medical Research Ethics Committee, faculty of medicine, Assiut University, Assiut, Egypt, and after obtaining written informed consents from all participating patients.

This prospective randomized clinical study will include ninety female patients with ASA I-II, aged 18-60 years, have BMI < 30 km\ m2 and scheduled for modified radical mastectomy with axillary dissection for management of breast cancer.

Excluded from the study are patients with known allergy to the study drugs, significant cardiac, respiratory, renal, CNS or hepatic disease, drug or alcohol abuse, pregnant women, patients refusing participation and psychiatric or mental illness that would interfere with perception and assessment of pain.

According to a random number sequence created by an internet web site (www.random.org), patients will be randomly assigned to three groups (30 patients each):

Group I: patients will receive oral lamotrigine 100 mg 1 hour before surgery with a sip of water.

Group II: patients will receive oral pregabalin 150 mg 1 hour before surgery with a sip of water.

Group III: patients will receive oral placebo 1 hour before surgery with a sip of water.

All patients preoperatively will be instructed in how to evaluate their own pain using NRS (numerical rating Scale) scored from Zero to ten where 0 = no pain and 10 = the worst pain imaginable for acute post-operative pain during the first 24 h after operation and LANSS (Leeds Assessment of Neuropathic Signs and Symptoms) Pain Scale at 3 and 6 months period after the surgery for chronic post-mastectomy pain assessment.

The LANSS pain scale is a simple bedside test used by the medical community to analyze and classify pain. It is a, conducted in two parts .i.e. a patient-completed questionnaire and a brief clinical assessment.

Its purpose is to assess whether the pain experienced is predominantly due to nerve damage or not. The LANSS scale is the only published tool with validity for discriminating between neuropathic and nociceptive pain, regardless if the disease-based diagnostic methods. It also assesses the severity of the pain or its causes.

It is composed of 7 items, five are symptom related and two are examination items.

1. Would you describe your pain as strange unpleasant sensations in your skin? (e.g. pricking, tingling, pins and needles) - Yes/No
2. Does the skin in the painful areas look different to normal? (e.g. mottled, more red/pink than usual) - Yes/No
3. Is the skin in the affected area abnormally sensitive to touch? (e.g. unpleasant sensations if lightly stroked, painful to wear tight clothes) - Yes/No
4. Does your pain come on suddenly in bursts for no apparent reason when you are still? (e.g. like electric shocks, 'bursting' or 'jumping' sensations) - Yes/No
5. Do you feel that skin temperature in the painful area has changed (e.g. hot, burning) - Yes/No
6. Does stroking the affected area of skin with a piece of cotton wool produce an unpleasant painful sensation? - Yes/No
7. Does touching the affected area of skin with a sharp needle feel sharper or duller when compared to an area of normal skin? - Yes/No Add values in parentheses for sensory description and examination findings to obtain overall score. TOTAL SCORE (maximum 24) If score < 12, neuropathic mechanisms are unlikely to be contributing to the patient's pain.

If score ≥ 12, neuropathic mechanisms are likely to be contributing to the patient's pain.

All patients from the 3 groups will not receive any pre-medications and the anesthetic technique will be standardized in all groups.

One hour before surgery, the patient will receive one of the study drugs with a sip of water. On admission to the operative room, patients will be connected to standard monitoring probes and an I.V. cannula will be inserted and a preload of 500 ml saline will be administered to all patients.

Pre-oxygenation for 3 minutes with 100% oxygen will be started. Anesthesia will be induced with 1.5-2 µg/kg fentanyl, 2-3 mg/kg propofol. Endotracheal intubation will be facilitated by cis-atracurium 0.15 mg/kg. Monitoring will include electoro-cardiography, non-invasive blood pressure, end tidal CO2 and SaO2. Anesthesia and muscle relaxation will be maintained by isoflurane 1-1.5 MAC in 50% oxygen/air mixture and cis-atracurium 0.03 mg/kg, respectively At the end of surgery, muscle relaxation will be reversed by neostagmine 0.5 µg/kg and atropine 0.02µg/kg. Patients will be extubated and transferred to the post-anesthesia care unit (PACU). In PACU the following data will be recorded: heart rate, mean arterial blood pressure, respiratory rate and oxygen saturation) at 0h (immediately postoperative), 2h, 4h, 6h, 12h and 24h post-operatively. NRS values at rest (NRS-R) and at movement (NRS-M) with abduction of ipsilateral arm will be also recorded at the same time points to evaluate acute postoperative pain.

Rescue post-operative analgesia in the form of I.V. Morphine through Patient controlled analgesia (PCA) with an initial bolus of 0.1 mg/ kg once pain is expressed followed by 1mg bolus upon pressing the button by the patient in pain with a lock-out interval of 15 minutes with no back-ground infusion. The time to first request of rescue analgesia and the total postoperative (24h) morphine consumption will be observed and recorded.

Postoperative adverse effects such as nausea, vomiting, skin rash, gastric upset and sedation will be recorded and treated. All patients will be scheduled for two visits into our pain clinic at the third and the sixth month postoperatively for assessment for the development of chronic post mastectomy pain using LANSS scale.

Our primary outcome measure is the total amount of rescue morphine received by patients for 24h postoperatively, secondary outcome measures include level of acute postoperative pain by NRS, the time to first request of rescue analgesia, development of chronic postmastectomy pain after 3 and 6 months postoperatively.

Sample size is calculated based on previous studies , assuming that a 20% reduction in postoperative morphine consumption would be clinically relevant , with α = 0.05 and the power of 0.8 , a samle size of 30 patient in each group will be necessary .

Analysis will perform using SPSS version 17 (Chicago-USA). Data will present as mean ± SD, numbers, frequencies, and percentages. ANOVA followed by post-hoc test willbe used for comparison of parametric data. Kruskal Wallis test will use to compare non-parametric data while Mann-Whitney will be used to compare between two groups. Chi-square test will be used for comparison between percentages and frequencies. P<0.05 will consider significant.

ELIGIBILITY:
Inclusion Criteria:

* female patients with ASA I-II, aged 18-60 years, have BMI < 30 km\ m2 and scheduled for modified radical mastectomy with axillary dissection for management of breast cancer

Exclusion Criteria:

- Excluded from the study are patients with known allergy to the study drugs, significant cardiac, respiratory , renal, CNS or hepatic disease, drug or alcohol abuse, pregnant women, patients refusing participation and psychiatric or mental illness that would interfere with perception and assessment of pain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Locations (1):
- Salma Komy, Asyut, Egypt

REFERENCES:
- [Background] Couceiro TC, Menezes TC, Valenca MM. Post-mastectomy pain syndrome: the magnitude of the problem. Rev Bras Anestesiol. 2009 May-Jun;59(3):358-65. doi: 10.1590/s0034-70942009000300012. English, Portuguese. PMID 19488550
- [Background] Maigaard S, Forman A, Andersson KE. Differences in contractile activation between human myometrium and intramyometrial arteries. Acta Physiol Scand. 1985 Jul;124(3):371-9. doi: 10.1111/j.1748-1716.1985.tb07672.x. PMID 3863453
- [Background] Panic A, Mijatovic D, Radosavac B. [The role of secondary prevention of alcoholism in the development of alcoholic epilepsy]. Med Pregl. 1986;39(9-10):445-8. No abstract available. Croatian. PMID 3587127
- [Background] Szabo AZ, Bocsan IC, Suciu S, Buzoianu AD. Comparative animal study of the antinociceptive efficacy of lamotrigine and gabapentin for the management of pain. Acta Physiol Hung. 2015 Dec;102(4):363-71. doi: 10.1556/036.102.2015.4.3. PMID 26690028
- [Background] Hunter JC, Gogas KR, Hedley LR, Jacobson LO, Kassotakis L, Thompson J, Fontana DJ. The effect of novel anti-epileptic drugs in rat experimental models of acute and chronic pain. Eur J Pharmacol. 1997 Apr 18;324(2-3):153-60. doi: 10.1016/s0014-2999(97)00070-8. PMID 9145766
- [Background] Taylor JC, Brauer S, Espir ML. Long-term treatment of trigeminal neuralgia with carbamazepine. Postgrad Med J. 1981 Jan;57(663):16-8. doi: 10.1136/pgmj.57.663.16. PMID 7279817
- [Background] Bertilsson L. Clinical pharmacokinetics of carbamazepine. Clin Pharmacokinet. 1978 Mar-Apr;3(2):128-43. doi: 10.2165/00003088-197803020-00003. PMID 346287
- [Background] Spina E, Pisani F, Perucca E. Clinically significant pharmacokinetic drug interactions with carbamazepine. An update. Clin Pharmacokinet. 1996 Sep;31(3):198-214. doi: 10.2165/00003088-199631030-00004. PMID 8877250
- [Background] Guay DR. Pregabalin in neuropathic pain: a more "pharmaceutically elegant" gabapentin? Am J Geriatr Pharmacother. 2005 Dec;3(4):274-87. PMID 16503325
- [Background] Frampton JE, Foster RH. Pregabalin: in the treatment of postherpetic neuralgia. Drugs. 2005;65(1):111-8; discussion 119-20. doi: 10.2165/00003495-200565010-00011. PMID 15610058
- [Background] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Background] Burke SM, Shorten GD. Perioperative pregabalin improves pain and functional outcomes 3 months after lumbar discectomy. Anesth Analg. 2010 Apr 1;110(4):1180-5. doi: 10.1213/ANE.0b013e3181cf949a. Epub 2010 Jan 26. PMID 20103545
- [Background] Buvanendran A, Kroin JS, Della Valle CJ, Kari M, Moric M, Tuman KJ. Perioperative oral pregabalin reduces chronic pain after total knee arthroplasty: a prospective, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):199-207. doi: 10.1213/ANE.0b013e3181c4273a. Epub 2009 Nov 12. PMID 19910619
- [Background] Rustagi A, Roychoudhury A, Bhutia O, Trikha A, Srivastava MV. Lamotrigine Versus Pregabalin in the Management of Refractory Trigeminal Neuralgia: A Randomized Open Label Crossover Trial. J Maxillofac Oral Surg. 2014 Dec;13(4):409-18. doi: 10.1007/s12663-013-0513-8. Epub 2013 May 24. PMID 26225004
- See also: Lamotrigine Versus Pregabalin in the Management of Refractory Trigeminal Neuralgia: A Randomized Open Label Crossover Trial. Ru — https://www.ncbi.nlm.nih.gov/pubmed/?term=26225004
- See also: Perioperative oral pregabalin reduces chronic pain after total knee arthroplasty: a prospective, randomized, controlled trial. — https://www.ncbi.nlm.nih.gov/pubmed/?term=19910619
- See also: Perioperative pregabalin improves pain and functional outcomes 3 months after lumbar discectomy. — https://www.ncbi.nlm.nih.gov/pubmed/?term=20103545
- See also: Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. — https://www.ncbi.nlm.nih.gov/pubmed/?term=18716003
- See also: Pregabalin: in the treatment of postherpetic neuralgia. — https://www.ncbi.nlm.nih.gov/pubmed/?term=15610058
- See also: Pregabalin in neuropathic pain: a more "pharmaceutically elegant" gabapentin — https://www.ncbi.nlm.nih.gov/pubmed/?term=16503325
- See also: Clinically significant pharmacokinetic drug interactions with carbamazepine — https://www.ncbi.nlm.nih.gov/pubmed/?term=8877250
- See also: Clinical pharmacokinetics of carbamazepine — https://www.ncbi.nlm.nih.gov/pubmed/?term=346287
- See also: Long-term treatment of trigeminal neuralgia with carbamazepine — https://www.ncbi.nlm.nih.gov/pubmed/?term=7279817
- See also: The effect of novel anti-epileptic drugs in rat experimental models of acute and chronic pain. — https://www.ncbi.nlm.nih.gov/pubmed/?term=9145766
- See also: Comparative animal study of the antinociceptive efficacy of lamotrigine and gabapentin for the management of pain — https://www.ncbi.nlm.nih.gov/pubmed/?term=26690028
- See also: Effects of preemptive analgesia with celecoxib or acetaminophen on postoperative pain relief following lower extremity orthopedic surgery — https://www.ncbi.nlm.nih.gov/pubmed/?term=23459777
- See also: A retrospective study of postmastectomy pain syndrome: incidence, characteristics, risk factors, and influence on quality of life — https://www.ncbi.nlm.nih.gov/pubmed/?term=24379736
- See also: Post-mastectomy pain syndrome: the magnitude of the problem — https://www.ncbi.nlm.nih.gov/pubmed/?term=19488550